CLINICAL TRIAL: NCT06861686
Title: A Modified Baveno Classification of Obstructive Sleep Apnoea Based on Sleepiness and Cardiovascular Scores: A Prospective Observational Cohort Study
Brief Title: A Modified Baveno Classification of Obstructive Sleep Apnoea Based on Sleepiness and Cardiovascular Scores
Status: Recruiting | Type: Observational
Sponsor: Wissenschaftliches Institut Bethanien e.V (Other)
Responsible Party: Sponsor
Other Study IDs: WI_24-1422
Record Dates: First submitted 2025-02-24; First posted 2025-03-06 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Obstructive Sleep Apnea (OSA)
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- weak treatment indication: Patients with obstructive sleep apnoea (OSA) for whom OSA-specific treatment is generally not recommended according to the Baveno classification
- intermediate treatment indication: Patients with obstructive sleep apnoea (OSA) for whom OSA-specific treatment should be considered based on individual assessment according to the Baveno classification
- strong treatment indication: Patients with obstructive sleep apnoea (OSA) for whom OSA-specific treatment is generally recommended according to the Baveno classification

SUMMARY:
The goal of this observational study is to evaluate a new classification system for obstructive sleep apnoea in patients with newly diagnosed obstructive sleep apnoea and monitor for long-term objective and subjective improvement.

ELIGIBILITY:
Inclusion criteria

1. Adult patient ≥40 years at the time of signed informed consent
2. Diagnosis of predominant obstructive sleep apnoea with a total apnoea-hypopnoea index of ≥5 /h based on a diagnostic sleep study (polysomnography or polygraphy, as per local standard). Predominant obstructive sleep apnoea defined as ≥70% of respiratory events classified as obstructive.
3. Signed and dated written informed consent in accordance with ICH-GCP and applicable local regulations

Exclusion criteria

1. >30% central respiratory events (apnoeas and hypopnoeas) within the diagnostic sleep study
2. Established sleep apnoea treatment within the last 12 months before study inclusion (positive airway pressure, mandibular advancement device, positional therapy)
3. Use, or need for chronic use, of any non-invasive positive pressure ventilation device
4. Participation in an interventional study and/or receiving investigational treatment(s)
5. Significant disease or condition, which, in the opinion of the investigator, may interfere with study procedures or cause concern regarding the patient's ability to participate in the study
6. Patients not expected to comply with the protocol requirements or not expected to complete the trial as scheduled (e.g. chronic alcohol or drug abuse or any other condition that, in the investigator's opinion, makes the patient an unreliable trial participant)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected obstructive sleep apnoea presenting for sleep medical evaluation
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in daytime sleepiness as measured by the Epworth Sleepiness Scale | From enrollment to the end of the individual observation period at 36 months
  The Epworth Sleepiness Scale total score ranges from 0-24. Higher values represent a larger extent of daytime sleepiness
Change in office systolic blood pressure | From enrollment to the end of the individual observation period at 36 months

SECONDARY OUTCOMES:
Change in office diastolic blood pressure | From enrollment to the end of the individual observation period at 36 months
Cardiovascular events (MACE) occurring after study inclusion, including but not limited to myocardial infarction, stroke, hospitalisation for cardiovascular-related treatment (e.g. heart failure, arrhythmia) | From enrollment to the end of the individual observation period at 36 months
Average OSA treatment usage | From enrollment to the end of the individual observation period at 36 months
  Average usage of the prescribed treatment for obstructive sleep apnea, measured as hours per day, derived from therapy device data
Number of patients who discontinue OSA treatment | From enrollment to the end of the individual observation period at 36 months
Change in Insomnia Severity Index total score | From enrollment to the end of the individual observation period at 36 months
  The Insomnia Severity Index (ISI) total score ranges from 0-28. Higher scores represent a larger extent of insomnia-related symptoms. Scores of 15 and above are indicative of clinical insomnia.
Change in subjective sleep length | From enrollment to the end of the individual observation period at 36 months
  Subjective sleep length as assessed via personal interview, measured in hours per night
Change in Fatigue Severity Scale mean score | From enrollment to the end of the individual observation period at 36 months
  The Fatigue Severity Scale (FSS) mean score ranges from 0-7, with higher values indicating a larger extent of fatigue.
Change in cognitive performance as assessed by the Montreal Cognitive Assessment (MoCA) total score | From enrollment to the end of the individual observation period at 36 months
  The Montreal Cognitive Assessment (MoCA) total score ranges from 0-30. A higher score represents a better cognitive performance. A result of 26 or higher is considered normal.
Change in average oxygen desaturation area as measured by overnight oximetry | From enrollment to the end of the individual observation period at 36 months
  The average oxygen desaturation area (unit: s*%) is automatically calculated from the oximetry signal of a single night poly(somno)graphy. Higher values indicate a larger extent of hypoxic burden.

CONTACTS AND LOCATIONS:
Overall Officials: Winfried J Randerath, Prof. Dr., Principal Investigator — Wissenschaftliches Institut Bethanien für Pneumologie e.V.
Locations (18):
- Belgium (2):
  - Antwerp University Hospital, Antwerp, Antwerp
  - UZ Leuven, Leuven, Vlaams-Brabant
- Centre Hospitalier Universitaire Grenoble Alpes, Grenoble, Isère, France
- Wissenschaftliches Institut Bethanien für Pneumologie e.V., Solingen, Germany
- Greece (4):
  - Department of Pulmonology, University General Hospital of Alexandroupolis, Medical School, Democritus University of Thrace, Alexandroupoli, Evros
  - Division of Pulmonology, Department of Clinical Therapeutics, National and Kapodistrian University of Athens, Medical School, Athens
  - University of Crete, Heraklion
  - Respiratory Failure Unit, G. Papanikolaou Hospital, Thessaloniki
- Italy (2):
  - Istituto Auxologico Italiano, Milan
  - Istituti Clinici Scientifici Maugeri IRCCS, Pavia
- Institute of Tuberculosis and Lung Diseases, Warsaw, Masovian Voivodeship, Poland
- Portugal (2):
  - Unidade Local de Saúde de Gaia e Espinho ULSGE - Unidade de Patologia do Sons, Vila Nova de Gaia, Porto District
  - Hospital Beatriz Ângelo, Unidade Local de Saúde Loures-Odivelas, Loures
- Romania (2):
  - Clinica Somnolog, Bucharest
  - University of Medicine and Pharmacy Dr. Victor Babes, Timișoara
- University Clinic of Respiratory and Allergic Diseases Golnik, Golnik, Slovenia
- Klinik für Pneumologie Universitätsspital Zürich, Zurich, Switzerland
- Ege University, Faculty of Medicine, Department of Respiratory Medicine, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided